CLINICAL TRIAL: NCT00151229
Title: Valsartan in Elderly Isolated Systolic Hypertension
Brief Title: Valsartan in Elderly Isolated Systolic Hypertension Study
Acronym: VALISH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VALISH study (Other)
Collaborators: Japan Cardiovascular Research Foundation (Other)
Responsible Party: Principal Investigator, Hiromi Rakugi, MD, PhD, Professor, Osaka University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAL-200310
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Aged; Systolic Hypertension
Keywords: isolated systolic hypertension; valsartan; target blood pressure
MeSH Terms: conditions — Isolated Systolic Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- strict control (Active Comparator): systolic blood pressure control: less than 140 mm Hg
  Interventions: Other: target blood pressure
- moderate control (Active Comparator): systolic blood pressure control: 140 mm Hg to 149 mm Hg
  Interventions: Other: target blood pressure

INTERVENTIONS:
Other: target blood pressure

SUMMARY:
The aim of this study is to compare the incidence of cardiovascular events between two target systolic blood pressure levels, below 140 mmHg and below 150 mmHg under treatment with valsartan in elderly isolated systolic hypertensive patients in Japan.

DETAILED DESCRIPTION:
Although antihypertensive therapy has been proven to reduce cardiovascular morbidity and mortality, it is unclear how much blood pressure should be decreased in elderly patients with hypertension. The Valsartan in Elderly Isolated Systolic Hypertension (VALISH) study is a multicenter parallel-group study comparing the incidence of cardiovascular events between two target systolic blood pressure levels, below 140 mmHg and below 150 mmHg, under treatment with valsartan, an angiotensin II receptor blocker, as an initial antihypertensive drug in elderly patients with isolated systolic hypertension. The number of patients to be recruited is 3,000 and the duration of follow-up is at least 2 years. This 3,000-patient trial was designed with a two-sided α level of 0.05 and 80% power to detect the difference in incidence of cardiovascular events between the target blood pressure levels based on estimation of the cardiovascular events ratio as 21.5/1,000 patient-years and 29.1/1,000 patient-years for the two blood pressure levels. The VALISH study, a large-scale investigator-initiated trial in Japan, will determine whether age should be considered in setting target blood pressure in treatment of isolated systolic hypertension in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged over 70 years and less than 85 years, regardless of sex.
* Patients with stable seated systolic blood pressure of over 160 mmHg and diastolic blood pressure of less than 90 mmHg at two visits within 2 to 4 weeks.
* Previously untreated patients or patients who are on other therapy that can be converted to valsartan.

Exclusion Criteria:

* Patients with secondary hypertension or malignant hypertension.
* Patients with seated systolic blood pressure of over 200 mmHg.
* Patients with seated diastolic blood pressure of over 90 mmHg.
* Patients with a history of cerebrovascular disorder or myocardial infarction within 6 months prior to enrolment in the study.
* Patients who underwent coronary arterioplasty within 6 months prior to enrolment in the study or patients who will undergo coronary arterioplasty within 6 months after entry.
* Patients with severe heart failure (NYHA functional classification III and IV).
* Patients with severe aortic stenosis or valvular disease.
* Patients with atrial fibrillation, atrial flutter, or serious arrhythmia.
* Patients with renal dysfunction with serum creatinine level of over 2 mg/dL.
* Patients with serious liver dysfunction.
* Patients with a history of hypersensitivity to valsartan.
* Other patients who are judged to be inappropriate for the study by the investigator or sub-investigator.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3079 (Actual)
Dates: Start 2003-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
composite cardiovascular events | participants will be followed for the duration of the study, an expected median follow-up 3.07 years
  sudden death, fatal or nonfatal stroke, fatal or nonfatal myocardial infarction, death because of heart failure, other cardiovascular death, unplanned hospitalization for cardiovascular disease, and renal dysfunction (doubling of serum creatinine to a level 2.0 mg per 100 mL or introduction of dialysis).

SECONDARY OUTCOMES:
sudden death | participants will be followed for the duration of the study, an expected median follow-up 3.07 years
stroke | participants will be followed for the duration of the study, an expected median follow-up 3.07 years
myocardial infarction | participants will be followed for the duration of the study, an expected median follow-up 3.07 years
heart failure | participants will be followed for the duration of the study, an expected median follow-up 3.07 years
hospitalization | participants will be followed for the duration of the study, an expected median follow-up 3.07 years
renal disorder | participants will be followed for the duration of the study, an expected median follow-up 3.07 years

CONTACTS AND LOCATIONS:
Overall Officials: Toshio Ogihara, MD, PhD, Principal Investigator — Department of Geriatric Medicine, Osaka University Graduate School of Medicine; Takao Saruta, MD, PhD, Principal Investigator — Department of Internal Medicine, Keio University School of Medicine
Locations (1):
- VALISH Data Center, ING Corporation, 8-21, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- [Background] Ogihara T, Saruta T, Matsuoka H, Shimamoto K, Fujita T, Shimada K, Imai Y, Nishigaki M. valsartan in elderly isolated systolic hypertension (VALISH) study: rationale and design. Hypertens Res. 2004 Sep;27(9):657-61. doi: 10.1291/hypres.27.657. PMID 15750259
- [Result] Ogihara T, Saruta T, Rakugi H, Matsuoka H, Shimamoto K, Shimada K, Imai Y, Kikuchi K, Ito S, Eto T, Kimura G, Imaizumi T, Takishita S, Ueshima H; Valsartan in Elderly Isolated Systolic Hypertension Study Group. Target blood pressure for treatment of isolated systolic hypertension in the elderly: valsartan in elderly isolated systolic hypertension study. Hypertension. 2010 Aug;56(2):196-202. doi: 10.1161/HYPERTENSIONAHA.109.146035. Epub 2010 Jun 7. PMID 20530299
- [Derived] Yano Y, Rakugi H, Bakris GL, Lloyd-Jones DM, Oparil S, Saruta T, Shimada K, Matsuoka H, Imai Y, Ogihara T. On-Treatment Blood Pressure and Cardiovascular Outcomes in Older Adults With Isolated Systolic Hypertension. Hypertension. 2017 Feb;69(2):220-227. doi: 10.1161/HYPERTENSIONAHA.116.08600. Epub 2017 Jan 3. PMID 28049699